CLINICAL TRIAL: NCT02181816
Title: Azilsartan/Amlodipine (Zacras) Combination Tablets LD & HD Specified Drug-use Survey "Long-term Use Survey"
Brief Title: Azilsartan/Amlodipine Combination Tablets LD & HD Specified Drug-use Survey "Long-term Use Survey"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 212-011; JapicCTI-142592 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azilsartan/Amlodipine: Azilsartan/Amlodipine combination tablets (20 mg/2.5 mg or 20 mg/5 mg), orally, once daily for up to 12 months. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Azilsartan/Amlodipine

INTERVENTIONS:
Drug: Azilsartan/Amlodipine — Azilsartan/Amlodipine combination tablets LD & HD
  Other Names: Zacras Combination Tablets LD & HD

SUMMARY:
The purpose of this survey is to evaluate the safety and efficacy of long-term use of azilsartan/amlodipine combination tablets Low Dose (LD) & High Dose (HD) (Zacras Combination Tablets LD & HD) in hypertensive patients in daily medical practice.

DETAILED DESCRIPTION:
This survey was designed to evaluate the safety and efficacy of long-term use of azilsartan/amlodipine combination tablets LD & HD (Zacras Combination Tablets LD & HD) in hypertensive patients in daily medical practice.

For adults, one azilsartan/amlodipine combination tablet (20 mg/2.5 mg [for LD tablets] or 20 mg/5 mg [for HD tablets] of azilsartan/amlodipine) is administered orally once daily. Azilsartan/amlodipine combination tablets should not be used as the first-line drug for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

-Hypertensive patients

Exclusion Criteria:

-Hypertensive patients who meet any of the following conditions, [1] to [3], are excluded from the survey:

1. Patients with a history of hypersensitivity to any of the ingredients of azilsartan/amlodipine combination tablets or other dihydropyridine drugs
2. Patients who are pregnant or having possibilities of being pregnant
3. Diabetic patients taking aliskiren fumarate (excluding those with markedly poor blood pressure control even after other antihypertensive treatment)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 271 investigative sites in Japan, from 26 June 2014 to 31 January 2017.
Pre-assignment Details: Participants with a historical diagnosis of hypertension were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Azilsartan/Amlodipine: Azilsartan/Amlodipine combination tablets (20 mg/2.5 mg or 20 mg/5 mg), orally, once daily for up to 12 months. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Azilsartan/Amlodipine
Started | 1090
Completed | 1031
Not Completed | 59
Not completed — Case Report Forms Uncollected | 38
Not completed — Protocol Deviation | 21

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Arm/Group | Azilsartan/Amlodipine
Number analyzed (Participants) | 1031
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482
  Male | 549
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 1031
Duration of Diagnosis of Hypertension [Count of Participants; unit: Participants] — Mean duration between start of study and first time of diagnosis of hypertension was reported.
  Participants
    < 1 Year | 167
    >= 1 Year and < 3 Years | 126
    >= 3 Years and < 5 Years | 63
    >= 5 Years | 312
    Unknown | 363
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 1027
    Inpatient | 4
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 909
    Had Predisposition to Hypersensitivity | 58
    Unknown | 64
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 245
    Had Medical Complications | 786
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 790
    Had Medical History | 164
    Unknown | 77
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 759
    (all) | 63.10 (14.601)
BMI [Mean (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height(m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/meter (m)^2
    number analyzed (Participants) | 709
    (all) | 24.92 (4.652)
Estimate Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliter (mL)/Minute (min)/1.73m^2] — Population: The number analyzed is the number of participants with data available for analysis.
  milliliter (mL)/Minute (min)/1.73m^2
    number analyzed (Participants) | 647
    (all) | 69.0 (19.64)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 489
  Current Smoker | 132
  Ex-Smoker | 195
  Unknown | 215
Drinking Habit [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 272
    No | 556
    Unknown | 203
Breast-Feeding [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 482
    Not Nursing | 479
    Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Events
Time Frame: Up to Month 12
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Azilsartan/Amlodipine
Number analyzed (Participants) | 1031
Percentage of Participants | 8.34

2. Secondary Outcome: Systolic Office Blood Pressure
Description: Systolic office blood pressure level at baseline, Month 1, and the final assessment point (up to Month 12) were reported.
Time Frame: Baseline, Month 1, and final assessment point (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had available efficacy data at baseline and post baseline. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury (mmHg)
Arm/Group | Azilsartan/Amlodipine
Number analyzed (Participants) | 1031
Millimeter of Mercury (mmHg)
  Baseline: number analyzed (Participants) | 1008
  Baseline | 149.5 (19.13)
  Month 1: number analyzed (Participants) | 833
  Month 1 | 137.2 (14.69)
  Final Assessment Point: number analyzed (Participants) | 1008
  Final Assessment Point | 133.0 (14.14)

3. Secondary Outcome: Diastolic Office Blood Pressure
Description: Diastolic office blood pressure level at baseline, Month 1, and the final assessment point (up to Month 12) were reported.
Time Frame: Baseline, Month 1, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan/Amlodipine
Number analyzed (Participants) | 1031
mmHg
  Baseline: number analyzed (Participants) | 1008
  Baseline | 83.3 (13.64)
  Month 1: number analyzed (Participants) | 833
  Month 1 | 77.4 (11.35)
  Final Assessment Point: number analyzed (Participants) | 1008
  Final Assessment Point | 75.0 (10.88)

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan/Amlodipine
All-Cause Mortality (participants affected / at risk) | 6/1031
Serious Adverse Events (participants affected / at risk) | 16/1031
Other Adverse Events (participants affected / at risk) | 15/1031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan/Amlodipine (N=1031)
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain stem haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Sudden death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Fall (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan/Amlodipine (N=1031)
Dizziness (Nervous system disorders) | 9
Blood creatinine increased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02181816/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT02181816/SAP_001.pdf